CLINICAL TRIAL: NCT01413685
Title: Interest of Calcineurin Activity for the Therapeutic Tacrolimus Monitoring in Renal Recipients
Brief Title: Calcineurin Activity in Renal Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no patient corresponding to criteria
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P071004
Record Dates: First submitted 2011-06-24; First posted 2011-08-10 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Renal Transplant Rejection
Keywords: tacrolimus; calcineurin; pharmacodynamic; TDM; pharmacokinetics
MeSH Terms: interventions — Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus (No Intervention): Determination of tacrolimus concentrations in whole blood and of calcineurin activities in lymphocytes at D8, D15, D21 (pharmacokinetics on 4 times samples), D28, M2 and M3 (residual measurement)
  Interventions: Other: Pharmacokinetics/dynamics

INTERVENTIONS:
Other: Pharmacokinetics/dynamics — Determination of tacrolimus concentrations in whole blood and of calcineurin activities in lymphocytes at D8, D15, D21 (pharmacokinetics on 4 times samples), D28, M2 and M3 (residual measurement)

SUMMARY:
The purpose is to define if calcineurin activity is a better biological parameter than blood concentration for the therapeutic tacrolimus monitoring.

DETAILED DESCRIPTION:
Some authors showed that the determination of calcineurin (enzyme of cyclosporin and tacrolimus action) activity was very interesting in bone narrow and hepatic transplant in order to monitor tacrolimus or cyclosporin. Indeed, Furthermore, target Tac concentrations still fail to provide in certain patients an appropriate immunosuppression reflected by rejection. Because a lack of data in renal transplant, we propose to study this population treated by tacrolimus, mycophenolate mofetil and corticoids in the first three months following the transplantation.

Our major aim is to study the relationship between calcineurin activity and immunologic events in 200 renal recipients treated with tacrolimus in the first three months following transplant. Immunologic events could be acute rejections and infraclinical rejections. The second aims are 1) if this relationship exists, to define the threshold predicting acute rejection using ROC-curve, 2) to define variations between pharmacodynamic (calcineurin activity) and pharmacokinetic (whole blood concentrations) tacrolimus monitoring and 3) to compare calcineurin activity in patients with acute rejection and those with borderline rejection. Blood samples will be collected into EDTA-containing vacutainers prior to the tacrolimus morning administration and at 2, 4, 6 and 9 hours following the administration at D7, D14 and D21. Whole blood tacrolimus concentrations and calcineurin activity were measured using LCMSMS and HPLC techniques. After D21, only residual measurements will be carried out at D28, M2 and M3. A comparative statistical analysis will be performed between data defined with and without rejection. In case of difference, a ROC curve analysis could define normal ranges of calcineurin activity.

This is the second study of the Sud FRANCILIEN Institute for Research in Nephrology-Transplantation defined with Nephrology departments in Mondor and BICETRE hospitals and the object "Interest of pharmacodynamics of immunosuppressive drugs in renal-transplant recipients" is a new theme of these teams.

ELIGIBILITY:
Inclusion Criteria:

* adult renal transplant recipients
* treated by tacrolimus (Prograf or ADVAGRAF), corticoids, Cellcept,

Exclusion Criteria:

* patients with a high risk of bad compliance (toxicomania, severe psychiatric troubles)
* multiorgan transplant patients with mTOR inhibitors treatments
* HIV infected patients
* lack of consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determination of tacrolimus concentrations in whole blood and of calcineurin activities in lymphocytes | at day 8, day15, day21 (pharmacokinetics on 4 times samples), day 28, month 2 and month 3 (residual measurement)

SECONDARY OUTCOMES:
Pharmacogenetics (3A5) | at day 8, day 15, day 21, day 28, month 2 and month 3
  * Genotyping of CYP3A5 * 3 (A6986G) and mdr-1: mutations of these proteins could explain the changes of absorption of tacrolimus.
  * For each patient, during the first month of treatment, 5 ml of blood will be collected on EDTA tube.
  * Genotyping is realized by the allelic discrimination technique Taqman, on a ABI Prism 7000 (TaqMan ®) in the Molecular Biology unit, Pharmacogenetics and Hormonology Bicêtre Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GRIMBERT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Henri Mondor, Créteil, France